CLINICAL TRIAL: NCT00086502
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of the Addition of MK0431 to Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Pioglitazone Therapy
Brief Title: Pioglitazone Add-on Study in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-019; Formally-A0604T2DPT; 2006_410
Record Dates: First submitted 2004-07-02; First posted 2004-07-05 (Estimated); Results first posted 2010-04-19 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sitagliptin 100 mg (Active Comparator): Sitagliptin 100 mg
  Interventions: Drug: Comparator: Sitagliptin; Drug: Comparator: Pioglitazone; Drug: Metformin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo; Drug: Comparator: Pioglitazone; Drug: Metformin

INTERVENTIONS:
Drug: Comparator: Sitagliptin — Sitagliptin 100 mg once daily, from Visit 4 through Visit 8. Day 1 through week 24
  Other Names: Januvia
  Arms: Sitagliptin 100 mg
Drug: Comparator: Placebo — Placebo (to match Sitagliptin 100 mg) once daily, from Visit 4 through Visit 8. Day 1 through Week 24
  Arms: Placebo
Drug: Comparator: Pioglitazone — Pioglitazone 30 mg or 45 mg once daily, Visit 2 through Visit 8
  Other Names: ACTOS
Drug: Metformin — Metformin rescue for patients meeting
  pre-specified glycemic criteria. Metformin 500 mg,once daily, Visit 4 through Visit 8

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an investigational drug in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patient has type 2 diabetes mellitus (T2DM)
* Patient is 18 years of age (or older)
* Patient is not pregnant or breast-feeding and does not plan to become pregnant for the duration of the study and poststudy follow-up period

Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or a history of ketoacidosis
* Patient required insulin within the prior 8 weeks
* Patient is on a weight loss program and is not in the maintenance phase
* Patient started on a weight loss medication (e.g., orlistat or sibutramine) within the prior 8 weeks
* Patient is on or likely to require treatment with treatment with immunosuppressive agents (e.g., cyclosporin, methotrexate)
* Patient has cirrhosis, active liver disease (other than fatty liver) or symptomatic gallbladder disease
* Patient has chronic myopathy, or a progressive neurological or neuromuscular disorder (e.g., multiple sclerosis or polymyositis)
* Patient has any of the following disorders within the past 6 months:

Acute coronary syndrome (e.g., MI or unstable angina), Coronary artery intervention, Stroke or transient ischemic neurological disorder.

* Patient has new or worsening signs or symptoms of coronary heart disease within the past 3 months
* Patient has severe peripheral vascular disease
* Patient has congestive heart failure
* Patient is HIV positive
* Patient has a clinically important hematological disorder (e.g., aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Patient has a history of neoplastic disease
* Patient has a history of alcohol or drug abuse within the past 3 years
* Patient has viral hepatitis (hepatitis B or C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2004-06; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Rosenstock J, Brazg R, Andryuk PJ, Lu K, Stein P; Sitagliptin Study 019 Group. Efficacy and safety of the dipeptidyl peptidase-4 inhibitor sitagliptin added to ongoing pioglitazone therapy in patients with type 2 diabetes: a 24-week, multicenter, randomized, double-blind, placebo-controlled, parallel-group study. Clin Ther. 2006 Oct;28(10):1556-68. doi: 10.1016/j.clinthera.2006.10.007. PMID 17157112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 15-Jul-2004.
  Last Patient Last Visit: 28-Sep-2005
  71 study centers worldwide
Pre-assignment Details: Patients ≥18 years of age with type 2 diabetes mellitus and inadequate glycemic control [hemoglobin A1C
  (HbA1c) ≥7.0 and ≤10.0%] who were on a stable dose of pioglitazone (≥30 mg/day) after a variable
  screening period were eligible to enter the 24-week study.
Groups:
- Sitagliptin 100 mg: The Sitagliptin 100 mg group includes data from patients randomized to receive treatment with 100 mg oral tablets of sitagliptin once daily (blinded) in addition to ongoing treatment with open-label pioglitazone 15 mg oral tablets (total daily dose 30 to 45 mg/day).
- Placebo: The Placebo group includes data from patients randomized to receive treatment with placebo matching sitagliptin 100 mg tablet once daily (blinded) in addition to ongoing treatment with open-label pioglitazone 15 mg oral tablets (total daily dose 30 to 45 mg/day).
Period: Overall Study
Arm/Group | Sitagliptin 100 mg | Placebo
Started | 175 | 178
Completed | 149 | 158
Not Completed | 26 | 20
Not completed — Adverse Event | 11 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Patient Moved | 1 | 1
Not completed — Protocol Discontinuation Criteria | 1 | 3
Not completed — Patient Accidentally Unblinded | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Placebo | Total
Number analyzed (Participants) | 175 | 178 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (10.4) | 56.9 (11.1) | 56.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 75 | 157
  Male | 93 | 103 | 196
Race/Ethnicity, Customized [Number; unit: participants]
  White | 127 | 129 | 256
  Black | 11 | 12 | 23
  Hispanic | 21 | 22 | 43
  Asian | 10 | 5 | 15
  Other | 6 | 10 | 16
HbA1c (Hemoglobin A1c) [Mean (Standard Deviation); unit: Percent] | 8.1 (0.8) | 8.0 (0.8) | 8.0 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Hemoglobin A1C) at Week 24
Description: HbA1c is measured as a percent. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Baseline and week 24
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. For FAS patients with no data at Week 24, the last non-baseline observed measurement was carried forward to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 163 | 174
Percent | -0.85 [-0.98 to -0.72] | -0.15 [-0.28 to -0.03]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Model terms: treatment; baseline; prior antihyperglycemic agent (AHA) therapy [not on AHA, monotherapy with oral AHA, peroxisome proliferator-activated receptor (PPAR)-based combination therapy]; Mean Difference (Net) = -0.70, 95% CI [-0.85 to -0.54], Standard Deviation 0.73

2. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Baseline and week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 163 | 174
mg/dL | -16.7 [-22.4 to -11.0] | 1.0 [-4.3 to 6.3]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -17.7, 95% CI [-24.3 to -11.0], Standard Deviation 30.9

ADVERSE EVENTS:
Time Frame: Week 0 through Week 24.
Description: Other (not including serious) adverse experience results represent those events included in the primary
  safety analysis for this study (i.e., events that occurred prior to the initiation of glycemic rescue therapy).
Arm/Group | Sitagliptin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 5/175 | 8/178
Other Adverse Events (participants affected / at risk) | 20/175 | 13/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=175) | Placebo (N=178)
Any Gastrointestinal Disorders (Gastrointestinal disorders) | 1 | 2
Ileitis (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0
Any General Disorders And Administration Site Conditions (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Any Hepatobiliary Disorders (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Any Immune System Disorders (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Any Injury, Poisoning And Procedural Complications (Injury, poisoning and procedural complications) | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Any Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Any Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Any Nervous System Disorders (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Any Pregnancy, Puerperium And Perinatal Conditions (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Any Psychiatric Disorders (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0
Any Skin And Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 1 | 0
Angioneurotic Oedema (Skin and subcutaneous tissue disorders) | 1 | 0
Any Vascular Disorders (Vascular disorders) | 0 | 1
Atherosclerosis Obliterans (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=175) | Placebo (N=178)
Any Infections And Infestations (Infections and infestations) | 11 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 11 | 6
Any Nervous System Disorders (Nervous system disorders) | 9 | 7
Headache (Nervous system disorders) | 9 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.